CLINICAL TRIAL: NCT06237452
Title: A Randomized, Double-Blind, Placebo-Controlled Phase 3 Study of VE303 for Prevention of Recurrent Clostridioides Difficile Infection
Brief Title: VE303 for Prevention of Recurrent Clostridioides Difficile Infection
Acronym: RESTORATiVE303
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Vedanta Biosciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: VE303-003
Record Dates: First submitted 2024-01-23; First posted 2024-02-01 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2025-10

CONDITIONS: Clostridium Difficile; Clostridium Difficile Infections; Clostridium Difficile Infection Recurrence; Clostridioides Difficile Infection; Clostridioides Difficile Infection Recurrence; CDI; C. Diff Infection; Recurrent Clostridium Difficile Infection; C.Difficile Diarrhea; Diarrhea Infectious
MeSH Terms: conditions — Clostridium Infections; Dysentery

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- VE303 (Experimental): Subjects assigned to the VE303 arm will take 3 capsules containing VE303 per day for 14 days after completing 10 to 21 days of standard of care antibiotic treatment for the qualifying CDI episode.
  Interventions: Biological: VE303
- Placebo (Placebo Comparator): Subjects assigned to the placebo arm will take 3 placebo capsules per day for 14 days after completing 10 to 21 days of standard of care antibiotic treatment for the qualifying CDI episode.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: VE303 — VE303 is a live biotherapeutic product (LBP) consisting of 8 clonally derived, nonpathogenic, nontoxigenic, commensal bacteria strains manufactured under Good Manufacturing Practices (GMP) conditions.
  Arms: VE303
Biological: Placebo — Placebo capsules contain microcrystalline cellulose. Placebo capsules are visually identical to and not discernible from VE303 capsules. Placebo capsules will not contain any VE303 drug product.
  Arms: Placebo

SUMMARY:
The overall objective of the RESTORATiVE303 study is to evaluate the safety and the Clostridioides difficile infection (CDI) recurrence rate at Week 8 in participants who receive a 14-day course of VE303 or matching placebo. The objectives and endpoints are identical for Stage 1 (recurrent CDI) and Stage 2 (high-risk primary CDI).

ELIGIBILITY:
Key Inclusion Criteria (For enrollment in Stage 1: recurrent CDI population):

* Age ≥ 12 years where permitted, and ≥ 18 years in other locations, with a laboratory-confirmed qualifying episode of CDI and at least 1 prior occurrence within the last 6 months

Key Inclusion Criteria (For enrollment in Stage 2: primary CDI with high-risk for recurrence population):

* Age ≥ 75 years with a laboratory-confirmed qualifying episode of CDI
* OR age ≥ 12 years where permitted, and ≥ 18 years in other locations, with least two of the following risk factors:

  1. Age ≥ 65 years
  2. Kidney dysfunction, defined as estimated creatinine clearance < 60 mL/min/1.73 m^2 at the time of the qualifying CDI episode
  3. History of regular use of a proton pump inhibitor (PPI) within the past 2 months and expectation of continued use of PPIs throughout the study
  4. History of a prior CDI episode between 6 and 12 months prior to enrollment
  5. Immunosuppression due to an underlying disease or its treatment
  6. Has undergone solid organ or hematopoietic stem cell transplantation

Key Inclusion Criteria (For enrollment in Stage 1 or 2):

* The qualifying episode of CDI must meet all the following criteria:

  1. New onset of ≥ 3 unformed bowel movements (ie, Types 5 to 7 on the Bristol stool scale) within 24 hours for 2 consecutive days
  2. CDI symptoms started within 4 weeks prior to initiation of standard of care (SoC) antibiotic therapy for CDI
  3. Stool sample collected before (or no later than 72 hours after) initiation of SoC antibiotic therapy that was positive in a CDI laboratory test, defined as enzyme immunoassay (EIA) for toxin A/B and glutamate dehydrogenase (GDH) with polymerase chain reaction (PCR) reflex testing for discordant EIA/GDH results, performed at either a local laboratory or the central laboratory
  4. Diarrhea considered unlikely to have another etiology
* Prior to receiving any study medication, the participant should:

  1. Receive and complete a course of SoC antibiotic therapy for at least 10 days, up to a maximum of 28 days (Note: choice of agent is at the physician's discretion and antibiotic tapering is not allowed). It is permissible for decentralized participants to be randomized during SoC antibiotic administration.
  2. Meet the criterion of a successful clinical response, defined attaining symptomatic control of the qualifying CDI episode, ie, < 3 loose/unformed bowel movements per 24 hours for at least 2 consecutive days
* Able to receive the first dose of study drug on the last planned day of SoC antibiotic administration for a qualifying CDI episode, or no later than 2 days after completion of antibiotic dosing
* Recovered from any complications of severe or fulminant CDI and be clinically stable by the time of randomization

Key Exclusion Criteria (For both Stage 1 and Stage 2):

* History of chronic diarrhea (defined as ≥ 3 loose stools per day lasting for at least 4 weeks) within 3 months prior to randomization that is not related to CDI
* Known or suspected toxic megacolon or small bowel ileus at the time of randomization
* History of confirmed celiac disease, inflammatory bowel disease, microscopic colitis, short gut, GI tract fistulas, or a recent episode (within 6 months of screening) of intestinal ischemia or ischemic colitis
* Receipt of bezlotoxumab during the course of SoC antibiotic treatment for the qualifying CDI episode
* Use of antidiarrheal drugs (eg, loperamide, diphenoxylate) within 3 days prior to the planned first dose of study drug
* Anticipated administration of oral or parenteral antibacterial therapy for a non-CDI indication after randomization through Week 24 (end of study)
* Probiotics, whether characterized as a dietary/food supplement, or a drug, are prohibited within 2 days before starting study drug and through the dosing period. (Note: consumption of food-based products such as yogurt, kombucha, and kefir are permitted.)
* Absolute neutrophil count (ANC) of < 0.5 ×10^9 cells/L on 2 consecutive occasions within 7 days prior to randomization, or sustained ANC < 1.0 × 10^9 cells/L

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 852 (Estimated)
Dates: Start 2024-05-20 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
CDI Recurrence Rate at Week 8 | 8 weeks
  Proportion of participants with laboratory-confirmed CDI recurrence before or at Week 8.

CONTACTS AND LOCATIONS:
Locations (202):
- United States (72):
  - Advanced Gastroenterology, P.C., Chandler, Arizona
  - Mayo Clinic Hospital, Phoenix, Arizona
  - Om Research, LLC, Apple Valley, California
  - Science 37 Inc (Remote/Home option), Culver City, California
  - Children's Hospital of Los Angeles, Los Angeles, California
  - VA San Diego Healthcare System, San Diego, California
  - North America Research Institute, San Dimas, California
  - Clinical Trials Management Services, Thousand Oaks, California
  - Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center, Torrance, California
  - Medical Research Center of Connecticut, Hamden, Connecticut
  - Hartford Hospital, Hartford, Connecticut
  - Gastro Florida, Clearwater, Florida
  - Proactive Clinical Research, LLC, Fort Lauderdale, Florida
  - Encore Borland-Groover Clinical Research, Jacksonville, Florida
  - GI Pros Research, Naples, Florida
  - Advanced Medical Research Center, Port Orange, Florida
  - KM International Research Operation LLC, Saint Cloud, Florida
  - James A. Haley Veterans' Hospital, Tampa, Florida
  - International Center for Research, Tampa, Florida
  - Summit Clinical Research, LLC, Athens, Georgia
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Metro Infectious Disease Consultants, Decatur, Georgia
  - Regional Infectious Diseases and Infusion Center, Inc., La Grange, Georgia
  - Gastrointestinal Specialists of Georgia, Marietta, Georgia
  - Snake River Research, PLLC, Idaho Falls, Idaho
  - Metro Infectious Disease Consultants, Burr Ridge, Illinois
  - NorthShore University Health System - Evanston Hospital, Evanston, Illinois
  - Innovative Clinical Research Center, LLC (ICRC), Island Lake, Illinois
  - Indiana University Health University Hospital, Indianapolis, Indiana
  - Deaconess GI Specialty Center, Newburgh, Indiana
  - University of Kansas Medical Center, Kansas City, Kansas
  - IDC Clinical Research, LLC, Wichita, Kansas
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - Johns Hopkins Hospital, Baltimore, Maryland
  - MGG Group Co., Inc., Chevy Chase Clinical Research, Chevy Chase, Maryland
  - Tufts Medical Center, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - LTC Charles S. Kettles VA Medical Center, Ann Arbor, Michigan
  - Henry Ford Health, Detroit, Michigan
  - Corewell Health William Beaumont University Hospital, Royal Oak, Michigan
  - University of Minnesota Medical Center, Minneapolis, Minnesota
  - MNGI Digestive Health, PA, Plymouth, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Delta Gastroenterology and Endoscopy Center, Southaven, Mississippi
  - University of Missouri, Columbia, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - St. Charles Clinical Research, Weldon Spring, Missouri
  - Rutgers Robert Wood Johnson Medical School, New Brunswick, New Jersey
  - South Jersey Infectious Disease, Somers Point, New Jersey
  - Northwell Health Division of Infectious Diseases, Manhasset, New York
  - NYU Grossman School of Medicine, New York, New York
  - New York Presbyterian Hospital, New York, New York
  - Manhattan Clinical Research, LLC, New York, New York
  - Syracuse VA Medical Center, Syracuse, New York
  - Montefiore Medical Center, The Bronx, New York
  - Toledo Institute of Clinical Research, Toledo, Ohio
  - Oklahoma City Veterans Affairs Healthcare System, Oklahoma City, Oklahoma
  - Susquehanna Research Group - Gastroenterology, Harrisburg, Pennsylvania
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Guthrie Medical Group, PC, Sayre, Pennsylvania
  - Frontier Clinical Research, Uniontown, Pennsylvania
  - Ralph H. Johnson VA Health Care System, Charleston, South Carolina
  - Lowcountry Infectious Diseases, P.A., Charleston, South Carolina
  - Medical University of South Carolina, Charleston, South Carolina
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - North Texas Infectious Disease Consultants, P.A., Dallas, Texas
  - University of Houston College of Pharmacy, Houston, Texas
  - BioStar Clinical Research, Katy, Texas
  - Simcare Medical Research, LLC, Sugar Land, Texas
  - Seattle Infectious Disease Clinic, Seattle, Washington
  - Virginia Mason Medical Center, Seattle, Washington
- Australia (4):
  - Concord Repatriation General Hospital, Concord, New South Wales
  - Westmead Hospital, Westmead, New South Wales
  - Monash Health, Clayton, Victoria
  - Melbourne Health, Parkville, Victoria
- Belgium (3):
  - Erasme University Hospital - Infectiology Department, Anderlecht
  - Universite Catholique De Louvain and Cliniques Universitaires Saint-Luc, Brussels
  - Universitair Ziekenhuis Gent, Ghent
- Brazil (7):
  - CCIH - Consultoria em Controle de Infecção Hospitalar Ltda, Belo Horizonte, Minas Gerais
  - Hospital Nossa Senhora das Graças, Curitiba, Paraná
  - CPCLIN - Centro de Estudos e Pesquisas em Molestias Infecciosas - Pesquisa Clínica, Natal, Rio Grande do Norte
  - Fundacao Universidade de Caxias do Sul - Hospital Geral de Caxias do Sul, Caxias do Sul, Rio Grande do Sul
  - Hospital de Clinicas de Porto Alegre - UFRGS, Porto Alegre, Rio Grande do Sul
  - Associação Educadora São Carlos AESC - Hospital Mãe de Deus - Centro de Pesquisa, Porto Alegre, Rio Grande do Sul
  - Hospital Alemao Oswaldo Cruz, São Paulo, São Paulo
- Bulgaria (6):
  - Medical Center Excelsior OOD, Base 1, Sofia, Sofia-Grad
  - UMHAT Burgas AD, Burgas
  - Multiprofile Hospital for Active Treatment St. Ivan Rilski Gorna Oriahovitsa EOOD, Gorna Oryahovitsa
  - Multiprofile Hospital for Active Treatment Sveti Nikolay Chuditvorets EOOD, Lom
  - Medicinski centar Hipokrat-N EOOD, Plovdiv
  - MHAT Dr.Ivan Seliminski - Sliven Ltd., Sliven
- Canada (12):
  - Alberta Health Services (AHS) - Foothills Medical Centre, Calgary, Alberta
  - University of Alberta, Edmonton, Alberta
  - CaRe Clinic, Red Deer, Alberta
  - Vancouver Coastal Health Research Institute Clinical Research Unit, Vancouver, British Columbia
  - The Moncton Hospital, Moncton, New Brunswick
  - NL Health Services, St. John's, Newfoundland and Labrador
  - Research St. Josephs Hamilton, Hamilton, Ontario
  - St. Joseph's Hospital - London, London, Ontario
  - Viable Clinical Research Corporation, Scarborough Village, Ontario
  - University Health Network, Toronto, Ontario
  - INTERMED groupe santé, Chicoutimi, Quebec
  - Centre Hospitalier de l Universite Laval (CHUL), Québec, Quebec
- Czechia (3):
  - Fakultni nemocnice Brno, Brno, Brno-město
  - Nemocnice Kyjov, p.o., Kyjov
  - Fakultni Nemocnice Ostrava, Ostrava-Poruba
- Aarhus University Hospital, Aarhus, Central Jutland, Denmark
- France (9):
  - Hospital St. Joseph, Les Paris, Auvergne-Rhône-Alpes
  - Hôpital du Bocage, Dijon, Franche-Comté
  - Centre Hospitalier Universitaire (CHU) de Reims - Hopital Robert Debre, Paris, Grand Est
  - CHU Bordeaux - Hopital Saint Andre Service de medecine interne et maladies infectieuses, Bordeaux Cedex, Hauts-de-France
  - Assistance Publique-Hopitaux de Paris (AP-HP) - Hopitaux Universitaires Paris Ile-de-France Ouest - Raymond-Poincare, Garches, Hauts-de-Seine
  - CHU de Nantes - Hôtel Dieu, Nantes, Loire-Atlantique
  - Assistance Publique Hôpitaux de Paris Hôpital Bichat- Claude Bernard - Département des maladies infectieuses et tropicales, Paris, Paris
  - Hôpital De La Croix Rousse - Gastroenterology, Lyon, Rhone
  - Chru De Tours, Tours
- Georgia (4):
  - ISR-GEO Med Res Clin Healthycore, Tbilisi, K'alak'i T'bilisi
  - LTD "Academician Vakhtang Bochorishvili Clinic", Tbilisi, K'alak'i T'bilisi
  - LTD "Aversi Clinic", Tbilisi, K'alak'i T'bilisi
  - LTD "Emergency Cardiology Center named by Acad.G.Chapidze", Tbilisi
- Germany (3):
  - University Hospital Frankfurt, Frankfurt am Main, Hesse
  - University Hospital Cologne AöR - Klinik I für Innere Medizin, Cologne, North Rhine-Westphalia
  - Epimed GmbH, Berlin, State of Berlin
- Hungary (5):
  - Bekes Varmegyei Kozponti Korhaz Dr. Rethy Pal Tagkorhaza, Békéscsaba, Bekes County
  - Szegedi Tudomanyegyetem Szent-Gyorgyi Albert Klinikai Kozpont, I. sz. Belgyogyaszati Klinika, Szeged, Csongrád megye
  - Komárom-Esztergom Vármegyei Szent Borbála Kórház, Tatabánya, Komárom-Esztergom
  - Semmelweis Egyetem, Budapest
  - Szabolcs-Szatmár-Bereg Vármegyei Oktatókórház Nyíregyházi Jósa András Tagkórház, Nyíregyháza
- Ireland (2):
  - Royal College of Surgeons in Ireland - Beaumont Hospital - Education and Research Centre, Dublin, Dublin
  - Our Lady of Lourdes Hospital, Drogheda, Louth
- Israel (9):
  - Rabin Medical Center - Beilinson Hospital, Petah Tikva, Central District
  - Tel Aviv Sourasky Medical Center, Tel Aviv, Central District
  - Shamir Medical Center (Assaf Harofeh), Ẕerifin, Central District
  - Carmel Medical Center, Haifa, Haifa District
  - Hillel Yaffe MC, Clinical Research Unit, Hadera, Haifa North
  - Hadassah Medical Centre, Jerusalem, Jerusalem
  - The Barzilai Medical Center, Ashkelon, Southern District
  - Rambam Health Care Campus, Haifa
  - The Chaim Sheba Medical Center, Tel Litwinsky
- Italy (11):
  - AO Nazionale SS. Antonio e Biagio e C. Arrigo, Alessandria, Alessandria
  - PO A. Manzoni di Lecco, ASST Lecco, Lecco, Lombardy
  - Ospedale Fatebenefratelli e Oftalmico, ASST Fatebenefratelli Sacco, Milan, Milano
  - Fondazione IRCCS San Gerardo dei Tintori, Monza, Monza E Brianza
  - Azienda Ospedaliera Universitaria Federico II, Napoli, Napoli
  - IRCCS Policlinico San Matteo, Università degli studi di Pavia, Pavia, Pavia
  - Azienda Ospedaliero-Universitaria di Modena, Policlinico di Modena - Malattie Infettive E Tropicali, Modena, Reggio Emilia
  - Osp. Pediatrico Bambino Gesù, IRCCS, Roma, Roma
  - Presidio Ospedaliero di Vittorio Veneto, Vittorio Veneto, Veneto
  - AOU Pisana - Stabilimento di Cisanello, Pisa
  - Ospedale Isola Tiberina Gemelli Isola, Roma
- Mexico (4):
  - Centro de Investigacion Medica Aguascalientes, Aguascalientes, Aguascalientes
  - Hospital Cardiologica Aguascalientes - Investigacion, Aguascalientes, Aguascalientes
  - Hospital Universitario "Dr. Jose Eleuterio Gonzalez" - Infectious Diseases, Monterrey, Nuevo León
  - FAICIC S de RL de C.V. - Gastroenterology, Veracruz, Veracruz
- Netherlands (2):
  - Leids Universitair Medisch Centrum (LUMC), Leiden, South Holland
  - Universitair Medisch Centrum (UMC) Utrecht - Julius Center for Health Sciences and Primary Care, Utrecht
- Poland (2):
  - NZOZ VIVAMED Jadwiga Miecz, Warsaw, Masovian Voivodeship
  - Gyncentrum sp. z o.o., Katowice, Silesian Voivodeship
- Portugal (7):
  - Unidade Local De Saude Do Alto Ave E.P.E., Guimarães, Braga District
  - Unidade Local De Saude De Coimbra E.P.E., Coimbra, Coimbra District
  - Unidade Local De Saude De Almada-Seixal E.P.E., Almada, Lisbon District
  - CCAB Centro Clinico Academico Braga Associacao - ULS Braga, Braga
  - Unidade Local de Saúde da Guarda (ULSG), Guarda
  - Unidade Local De Saude De Santo Antonio E.P.E., Porto
  - Unidade Local De Saude De Gaia/Espinho E.P.E., Vila Nova de Gaia
- Romania (6):
  - Institutul de Boli Infecțioase Prof Dr Matei Bals - Infectious diseases V, Bucharest, București
  - Spitalul Clinic de Boli Infectioase si Tropicale Dr Victor Babes, Bucharest, București
  - Spitalul Clinic de Boli Infectioase Cluj-Napoca, Cluj-Napoca, Cluj
  - Centrul Medical Renasterea, Craiova, Dolj
  - Spitalul Clinic de Boli Infectioase Sfanta Parascheva Iasi - Infectious diseases I, Iași, Iaşi
  - Spitalul Clinic Judetean De Urgenta Pius Brinzeu Timisoara, Timișoara, Timiș County
- South Korea (4):
  - Yonsei University, Wonju Severance Christian Hospital, Wŏnju, Gangwon-do
  - Samsung Medical Center, Seoul, Seoul Teugbyeolsi
  - The Catholic University of Korea, Seoul St. Mary's Hospital, Seoul, Seoul Teugbyeolsi
  - Hallym University Kangnam Sacred Heart Hospital, Seoul, Seoul Teugbyeolsi
- Spain (15):
  - Hospital Universitari Germans Trias i Pujol, Badalona, Barcelona
  - Hospital Universitario de Bellvitge, Barcelona, Barcelona
  - Hospital Universitario Mutua de Terrassa, Terrassa, Barcelona
  - H. U. Donostia, San Sebastián, Guipúzcoa
  - Gregorio Marañón University Hospital, Madrid, Madrid
  - Hospital Universitario La Paz - UCICEC, Madrid, Madrid
  - Hospital Universitario Puerta De Hierro Majadahonda, Majadahonda, Madrid
  - Hospital Universitario Virgen Macarena, Seville, Sevilla
  - Complexo Hospitalario Universitario A Coruña, A Coruña
  - Hospital General Universitario Dr Balmis, Alicante
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital de La Santa Creu i Sant Pau, Barcelona
  - Hospital Universitario Reina Sofia, Córdoba
  - Hospital Universitario Ramón y Cajal, Madrid
  - Hospital Universitario Virgen De La Macarena, Seville
- Taiwan (3):
  - KMU Chung-Ho Memorial Hospital, Kaohsiung City, Kaohsiung
  - China Medical University Hospital - Infectious, Taichung, Taichung
  - Chang Gung Medical Foundation - LinKou Chang Gung Memorial Hospital, Taoyuan District, Taoyuan
- United Kingdom (8):
  - Royal Devon University Healthcare NHS Trust, Exeter, Devon
  - The Royal Bournemouth Hospital, Bournemouth
  - North Bristol NHS Trust - Southmead Hospital, Clinical Research Centre, Bristol
  - NHS Lothian - Western General Hospital, Edinburgh
  - Royal Free London NHS Foundation Trust, London
  - St.Thomas' Hospital, London
  - Northern General Hospital, Sheffield
  - Morriston Hospital, Swansea

REFERENCES:
- See also: At-home study participation for US participants - Science 37 — https://studies.science37.com/s37/inf-dis/?utm_source=peggylillisfoundation&utm_medium=advocacy&utm_campaign=cdiff_PLF
- See also: US Participants - Determine if you qualify — https://restorative303study.com/?utm_source=clinicaltrialsgov&utm_medium=referral